CLINICAL TRIAL: NCT06468865
Title: Continuous Glucose Monitoring in Treatment of Postprandial Hypoglycemia After Gastric Bypass Surgery: The HypoSurge Randomized Clinical Trial
Brief Title: Glucose Monitoring in Treatment of Postprandial Hypoglycemia After Gastric Bypass Surgery
Acronym: HypoSurge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Heidi Borgeraas, Principal investigator, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 596343
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Hypoglycemia Non-Diabetic; Gastric Bypass Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous glucose monitor (Experimental): The participants will wear a blinded (i.e. glucose levels are not displayed) Dexcom® G7 continuous glucose monitor for one week during the screening week.
  After the screening week, the patients will be given dietary guidance on how to avoid hypoglycaemia and be given a capillary glucometer (standard treatment procedure). The patients will also use a continuous glucose monitor and receiver which displays real-time glucose levels, for 6 weeks, to learn how to avoid hypoglycaemia.
  Interventions: Device: Continuous glucose monitor (Dexcom® G7)
- No continuous glucose monitor (No Intervention): The participants will wear a blinded (i.e. glucose levels are not displayed) Dexcom® G7 continuous glucose monitor for one week during the screening week.
  After the screening week, the patients will be given dietary guidance on how to avoid hypoglycaemia and be given a capillary glucometer (standard treatment procedure). The patients will not use a continuous glucose monitor during the following 5 weeks, but during week 6 the patient will wear a blinded continuous glucose monitor.

INTERVENTIONS:
Device: Continuous glucose monitor (Dexcom® G7) — Continuous glucose monitors measures glucose levels in the interstitial fluid every 5 minutes
  Arms: Continuous glucose monitor

SUMMARY:
The goal of this clinical trial is to learn if continuous glucose monitoring works to treat postprandial hypoglycaemia in patients who have undergone gastric bypass surgery. The main question it aims to answer is:

• Is continuous glucose monitoring superior to usual care for prevention of postprandial hypoglycaemia in patients with verified postprandial hypoglycaemia after gastric bypass surgery?

Researchers will compare continuous glucose monitoring to usual care to see if continuous glucose monitoring works to treat postprandial hypoglycaemia.

Participants will:

* Use a continuous glucose monitor for 6 weeks or use no continuous glucose monitor for 5 weeks and wear a blinded continuous glucose monitor for 1 week.
* Visit the clinic 2-3 times and have 2-3 phone consultations.
* Register symptoms of hypoglycaemia, answer questionnaires, undergo a 24-hour dietary recall interview conducted by a registered dietitian, measure weight and body composition and take blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Gastric bypass surgery at least 1 year ago
* Age ≥18 years
* Symptomatic postprandial hypoglycaemia; capillary glucose level <3.0 mmol/L 1-4 hours after meals

Exclusion Criteria:

* Not able to give informed consent
* Reduced compliance due to severe mental and psychiatric conditions
* Use of insulin or sulfonylureas
* Use of systemic corticosteroids
* Primary or secondary adrenal insufficiency
* Insulinoma
* Severe heart-, lung, liver- or kidney disease, cancer, malnutrition and other medical conditions causing fragility
* Performed bariatric revisional surgery
* Drug- or alcohol abuse
* Pregnancy
* Use of acarbose or octreotide in the treatment of postprandial hypoglycemia
* Use of continuous glucose monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
• Difference between the two treatment arms in change in weekly diurnal time spent with hypoglycaemia (interstitial glucose <3.0 mmol/L) from the screening week to week 6, measured with a continuous glucose monitor. | Screening (week 0) and week 6
  Interstitial glucose is measured for one week during the screening week and for one week during week 6.

SECONDARY OUTCOMES:
• Difference between the two treatment arms in change in weekly diurnal time spent with hypoglycaemia (interstitial glucose <3.9 mmol/L) from the screening week to week 6, measured with a continuous glucose monitor. | Screening (week 0) and week 6
  Interstitial glucose is measured for one week during the screening week and one week during week 6.
• Difference between the two treatment arms in change in weekly time (total and nocturnal) spent with hypoglycaemia (interstitial glucose <3.0 mmol/L and <3.9 mmol/L) from the screening week to week 6, measured with a continuous glucose monitor. | Screening (week 0) and week 6
  Interstitial glucose is measured for one week during the screening week and one week during week 6.
• Difference between the two treatment arms in change in weekly events (diurnal, total and nocturnal) of hypoglycaemia (interstitial glucose <3.0 mmol/L and <3.9 mmol/L) from the sceening week to week 6, measured with a continuous glucose monitor. | Screening (week 0) and week 6
  Interstitial glucose is measured for one week during the screening week and one week during week 6.

CONTACTS AND LOCATIONS:
Locations (1):
- 1Department of Endocrinology, Obesity and Nutrition, Vestfold Hospital Trust, Tønsberg, Vestfold, Norway